CLINICAL TRIAL: NCT01454466
Title: Partial Posterior Hyaloidectomy in Macular Surgery : A Modified Procedure of Vitrectomy to Prevent Retinal Break Related to Induction of a Posterior Vitreous Detachment
Brief Title: Partial Posterior Hyaloidectomy in Macular Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011-05-011
Record Dates: First submitted 2011-10-17; First posted 2011-10-19 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Retinal Break; Retinal Detachment
Keywords: prevention; retinal break; vitrectomy; partial posterior hyaloidectomy
MeSH Terms: conditions — Retinal Perforations; Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Partial posterior hyaloidectomy (a modified procedure of vitrectomy) — The core vitrectomy entails more extensive removal of vitreous gel, in contrast to the conventional core vitrectomy. IPVD was conducted by engaging the attached posterior cortical vitreous with a 23-gauge needle with angulated tip in the area adjacent to the optic disc followed by gently moving the tip to approximately 3 disc diameters away from the margin of the optic disc. After then, slightly elevating the tip in a posteroanterior direction with slowly proceeding it to the extent that we planned. With IPVD, the surgeon was able to visualize a floating Weiss ring in all of the cases. Active suction to initiate IPVD was not used in any of the cases. In the temporal direction, the extension of a PVD was restricted to approximately 2 disc diameters distance beyond the margin of temporal major vascular arcade

SUMMARY:
To evaluate the effect of partial posterior hyaloidectomy on preventing iatrogenic retinal breaks related to induction of a posterior vitreous detachment

DETAILED DESCRIPTION:
The induction of a posterior vitreous detachment (IPVD) during vitrectomy have been suggested as one of the etiologies of iatrogenic retinal break related to vitrectomy.The iatrogenic retinal breaks related to IPVD usually develop near or anterior to the equatorial region.

Thus, the investigators hypothesized that this complication could be prevented by restricting the extent of IPVD, and planned a modified procedure of vitrectomy in which the extent of IPVD and removal of vitreous cortex was restricted to about slightly beyond the margin of temporal major vascular arcade.

The investigators have termed this procedure, partial posterior hyaloidectomy. Unlike RRD or proliferative diabetic retinopathy, lesions are localized within the major vascular arcade in macular disorders so that macular disorders could be an eligible indication for this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Cases of idiopathic ERM or idiopathic MH without evidence of PVD preoperatively

Exclusion Criteria:

* history of previous intraocular surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
incidence of intraoperative and postoperative retinal break related to surgery | postoperative 3 to 6 months
  The eyes that completed a follow-up of at least 3 months were included in the result analysis. The incidence of retinal breaks related to the surgery was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Se Woong Kang, M.D., Study Chair — Samsung Medical Center; Jae Hui Kim, M.D., Principal Investigator — Samsung Medical Center